CLINICAL TRIAL: NCT05460884
Title: Investigating the Effects of Seaweed Extract on Blood Glucose and Insulin Levels After a Meal in Healthy Subjects
Brief Title: Effects of Seaweed Extract on Postprandial Response to White Bread
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Akristic, Assistant Professor, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: LS-19-84
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Glycemic Control; Diabetes Mellitus Risk; Glucose Intolerance; Postprandial Hyperglycemia; Healthy Subjects
Keywords: seaweed; Ascophyllum; blood glucose; insulin; postprandial; hyperglycemia
MeSH Terms: conditions — Glucose Intolerance; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: physically incorporated in the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): Participants will consume 109 g of white bread
  Interventions: Dietary Supplement: White bread
- Experimental 1: Seaweed extract at lower dose (LD) and white bread (Experimental): Participants will consume 109 g of white bread with 0.5g of seaweed extract
  Interventions: Dietary Supplement: Seaweed extract LD and white bread
- Experimental 2: Seaweed extract at higher dose (HD) and white bread (Experimental): Participants will consume 109 g of white bread with 1g of seaweed extract
  Interventions: Dietary Supplement: Seaweed extract HD and white bread

INTERVENTIONS:
Dietary Supplement: Seaweed extract LD and white bread — 109g of white bread with 0.5g of seaweed extract
  Arms: Experimental 1: Seaweed extract at lower dose (LD) and white bread
Dietary Supplement: Seaweed extract HD and white bread — 109g of white bread with 1g of seaweed extract
  Arms: Experimental 2: Seaweed extract at higher dose (HD) and white bread
Dietary Supplement: White bread — 109g of white bread
  Arms: Control

SUMMARY:
The study is designed to determine whether seaweed extract added to a carbohydrate-rich meal, can lower blood glucose levels after its consumption, and hence lower its glycaemic index, and if this effect is mediated through effects on insulin. It is designed as an acute, randomised, cross-over, controlled, three-arm dietary intervention trial in healthy subjects. Participants will be asked to consume either white bread, white bread with lower dose of seaweed extract or white bread with higher dose of seaweed extract.The effects on plasma glucose levels and levels of insulin will be determined over 3 hours after the consumption.

DETAILED DESCRIPTION:
It has been shown in a large number of in vitro studies that seaweed extracts act as potent inhibitors of enzymes of carbohydrate digestion suggesting their potential to modulate postprandial glycaemic response and prevent the damaging effects of hyperglycaemic state. However, the results from human trials are limited and inconsistent.

The investigators confirmed that the in vitro inhibitory effects of seaweed extracts depend on the type, level and ratio of bioactive compounds, and optimised the composition of the extract to obtain the most potent one, to be tested in the proposed study.

The present study will determine whether the seaweed extract added to a carbohydrate-rich meal, can lower blood glucose levels after its consumption, and hence lower its glycaemic index, and if this effect is mediated through effects on insulin or determined by the individual levels of digestive enzymes.

Healthy volunteers will be asked to consume three different meals: (1) white bread; (2) white bread with the lower dose (LD) of the extract; (3) white bread with the higher dose (HD) of the extract

The levels of glucose and insulin will be measured in plasma isolated from blood samples obtained before and up to 3 hours after the consumption of each meal.

Additional measurements taken at the screening will include blood pressure values and blood lipids levels. All participants will be characterized for the activity of salivary a-amylase.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Healthy

Exclusion Criteria:

* Smoking
* Diagnosis of any chronic illness (including diabetes, hypertension, gastrointestinal diseases etc.)
* On long term prescribed medication (except contraceptives)
* Pregnant or lactating
* On a special diet or dietary regimen (for weight management or if regularly consuming fruit extract supplements)
* Allergy to fruits vegetables or pollen
* Unwillingness to follow dietary recommendations or record the diet during recommended period
* Donated blood 4 weeks before or intend to donate blood during the study or 4 weeks after the last study samples
* Participation in another research project in parallel which also involves dietary intervention (e.g. taking vitamin supplements) or requires sampling of blood

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-12 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in maximal incremental plasma glucose level (iCmax) between baseline and endpoint within intervention groups vs. control. | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min
  The incremental glucose levels will be determined for each time point (at 15, 30, 45, 60, 90, 120, 150 and 180 min) as the change in plasma glucose levels after the consumption of both levels of seaweed extracts concomitantly with white bread, or white bread only, compared to the glucose levels before the consumption of test meals (baseline value, t=0min).

SECONDARY OUTCOMES:
Changes in area under the curve of incremental plasma glucose levels (iAUC) in the intervention group vs. control | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min
  The glucose iAUC will be determined from all incremental plasma glucose levels at the defined time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 min) after the consumption of test and control meals based on trapezoid rule.
Changes in plasma insulin levels between baseline and endpoint within the intervention group vs. control | Baseline, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min
  nsulin levels measured at the baseline and at each time point (at 15, 30, 45, 60, 90,120, 150 and 180 min) after the consumption of test and control meals.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food and Health Volunteer Suite; Science Center South, UCD, Dublin, Dublin 2, Ireland

IPD SHARING:
Plan to Share IPD: No
Data will be archived in an anonymised form. Following completion of the study the data will only be accessible by the PIs. Access to the data by a 3rd party will only be given through collaboration with one of the existing PIs. The data may be shared for other research projects, and in an anonymised form. Consent to share the data for such purposes is requested in the study consent form.